CLINICAL TRIAL: NCT03522896
Title: Effect of Hesperidin in Orange Juice on Glycemic Response in Healthy Volunteers
Brief Title: Effect of Orange Juice on Glycemic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Gary Williamson, Prof, University of Leeds
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: MEEC15-044b
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Effect of Food on Postprandial Hyperglycemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control meal (Placebo Comparator): glucose, fructose, sucrose, malic acid and citric acid in water
  Interventions: Other: control
- test meal 1 (Experimental): orange juice with added hesperidin (low dose)
  Interventions: Other: test meal 1
- test meal 2 (Experimental): orange juice with added hesperidin (high dose)
  Interventions: Other: test meal 2
- test meal 3 (Experimental): diluted orange juice with added hesperidin
  Interventions: Other: test meal 3

INTERVENTIONS:
Other: control — balancing sugars and organic acids
  Arms: control meal
Other: test meal 1 — orange juice plus hesperidin low dose
  Arms: test meal 1
Other: test meal 2 — orange juice plus hesperidin higher dose
  Arms: test meal 2
Other: test meal 3 — diluted orange juice plus hesperidin low dose
  Arms: test meal 3

SUMMARY:
Orange juice naturally contains high concentrations of hesperidin, which affects glucose absorption in in vitro experiments. This study is to test if hesperidin and other components of orange juice (not other sugars or organic acids) affect the post-prandial blood glucose concentration derived from sugars already present in the orange juice.

DETAILED DESCRIPTION:
Healthy volunteers will consume orange juice with added water or food-grade hesperidin.

ELIGIBILITY:
Inclusion Criteria:

* fasting blood glucose below 5.9 mM

Exclusion Criteria:

* fasting glucose above 6 mM pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

PRIMARY OUTCOMES:
Blood glucose concentration | 3 hours
  iAUC/[glucose]max

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leeds, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided